CLINICAL TRIAL: NCT06626698
Title: Effect of Electrical Muscle Elongation vs. Static Stretching in the Leg Muscles Contracture
Brief Title: Electrical Stimulation vs. Static Stretching in the Leg Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Aurora Castro Mendez, Principal Investigator. Aurora Castro-Méndez., University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US-elect26
Record Dates: First submitted 2024-09-23; First posted 2024-10-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Muscle Fatigue
Keywords: Achilles tendon; gastrocnemius muscle; electric stimulation; static stretching; articular Range of Motion; randomized Clinical trial; Longitudinal; muscle shortening; Session duration; Comparision group; Electric muscle elongation; triceps surae
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the Experimental Group (Electrical Muscle Elongation, EME) or the Control Group (Static Stretching, SS) to compare the immediate and short-term effects of the interventions.
Who Masked: Participant
Masking Description: This was a single-blind study. The Participants were blinded to the specific intervention they received, as both the Electrical Muscle Elongation (EME) technique and the Static Stretching (SS) technique involved similar positioning and physical manipulation of the ankle, making it challenging for them to distinguish the exact treatment modality.
  However, the Investigator (A.C-M, responsible for allocation and data recording) and the Care Provider (L.R-F, the podiatrist who applied the corresponding technique) were not blinded to the group assignment due to the distinct nature of the two interventions (one involving electrotherapy equipment and the other not).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: static stretching (Experimental): Passive static stretching of the posterior leg muscles. Single session of 30 seconds per 4 sets with 30 seconds of rest
  Interventions: Other: Static stretching
- Experimental: EME (Experimental): Electrical muscle elongation with interferential current. Dosage: 4kHz frequency and 100Hz frequency modulation amplitude. Self-adhesive surface electrodes (50x90 mm) and SONOPULS-492 equipment. Single session of 30 seconds per 4 sets with 30 seconds of rest.
  Interventions: Device: Electrical muscle elongation

INTERVENTIONS:
Other: Static stretching — A passive static stretch of the posterior leg muscles will be performed with the subject in a supine position and knees extended, starting with the ankle at 90º and continuing until reaching the maximum tolerated dorsiflexion.
  Arms: Experimental: static stretching
Device: Electrical muscle elongation — The intervention will be performed with the subject in a supine position with knees extended. Electrodes will be placed on the gastrocnemius muscles of the leg being assessed. The parameters will be selected. Static stretching will begin until resistance is felt, at which point the intensity of the electrical current will be increased to induce a visible and tolerable contraction. Simultaneously, the subject will be asked to perform an isometric contraction of the antagonist muscles, resisted by the investigator. When the subject feels the stretch again, the intensity of the current will be increased once more until a new movement barrier is reached.
  Arms: Experimental: EME

SUMMARY:
The retraction of the posterior leg muscles consists of a shortening of the muscle fibers that limits ankle dorsiflexion. The objective of this randomized controlled clinical trial (RCT) with a double-blind technique and longitudinal chronology is to evaluate the short-term effect of electrostimulation associated with muscle stretching (electrical muscle elongation technique or EME) compared to static stretching in adult subjects with shortening of the posterior leg muscles.

The main questions it seeks to answer are:

* Are there significant differences in the short-term effect of electrical muscle elongation versus static stretching exercises on the gastrocnemius complex and Achilles tendon in young adults?
* Does the ankle's range of motion increase in both weight-bearing and non-weight-bearing positions?
* Does muscle strength increase in ankle plantar flexion?

The researchers will compare the group receiving electrical muscle elongation with interferential current to the group receiving passive static stretching to assess whether there are significant differences in the effects on the ankle's range of motion and the muscle strength of the posterior leg muscles.

Participants in this study will perform the following tasks:

* Receive a session of electrical muscle elongation with TENS and static stretching performed by the researcher.
* Follow the instructions during the intervention.
* Undergo evaluations of ankle range of motion and plantar flexor muscle strength
* Record their level of satisfaction after the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects affiliated with or related to the University of Seville.
* Those with muscular shortening of the posterior chain of the limb.

Exclusion Criteria:

* Subjects who engage in sports activity above the average of the sample or who follow an organized stretching program for the posterior leg muscles.
* Hyperlaxity
* History of musculoskeletal, neuromuscular injuries, joint disease, surgery on the lower leg, or serious illness.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the ankle range motion | Through study completion, an average of 2 weeks.
  Assessment will be conducted in a prone position using a two-arm goniometer with the knee flexed and extended, as well as in a standing position with a digital inclinometer with the knee flexed and extended. Additionally, the distance from the big toe to the wall will be measured with a tape measure. This evaluation is carried , before and after a electric stimulation to compare if this measure may be different after this intervention At the beginning, during the intervention and a week later.
leg muscular force | Through study completion, an average of 2 weeks.
  Assessment will be conducted with the subject in a supine position and with knees extended. The plantarflexor strength of the ankle will be measured using a portable dynamometer. Three measurements will be taken, and the average will be calculated. this measure is carried on to evaluation if the force of the posterior leg muscles may be increased At the beginning, during the intervention and a week later.

SECONDARY OUTCOMES:
Patient Global Impression of Improvement cuestionarie | At the end of the study, an average of 2 weeks
  A questionnaire indicating the global impression of improvement after the intervention will be administered at the end of the study. It is to assesment is this study it is confortable for the patient The scale has a total score from 1 to 7. A value of 1 indicates great improvement and a value of 7 indicates that the patient is very unwell.

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Castro PhD, Principal Investigator — University of Seville
Locations (1):
- Área Clínica de Podología, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mizuno T. Combined Effects of Static Stretching and Electrical Stimulation on Joint Range of Motion and Muscle Strength. J Strength Cond Res. 2019 Oct;33(10):2694-2703. doi: 10.1519/JSC.0000000000002260. PMID 29023326
- [Result] Espejo-Antunez L, Lopez-Minarro PA, Garrido-Ardila EM, Castillo-Lozano R, Dominguez-Vera P, Maya-Martin J, Albornoz-Cabello M. A comparison of acute effects between Kinesio tape and electrical muscle elongation in hamstring extensibility. J Back Musculoskelet Rehabil. 2015;28(1):93-100. doi: 10.3233/BMR-140496. PMID 25061028
- [Result] Espejo-Antúnez L, López-Miñarro PA, Albornoz-Cabello M, Garrido-Ardila EM. Acute effect of electrical muscle elongation and static stretching in hamstring muscle extensibility. Science & Sports. 1 de febrero de 2016;31(1):e1-7.
- [Result] Espejo Antúnez L, Maya Martín J, Cardero Durán MA, Albornoz Cabello M. Aumento de la extensibilidad isquiotibial tras aplicar elongación muscular eléctrica. Fisioterapia. 1 de mayo de 2012;34(3):112-7.